CLINICAL TRIAL: NCT05563974
Title: Feasibility and Acceptability of a Family-led Care Model to Increase Coverage and Quality of Postnatal Care in Ethiopia
Brief Title: Family Led Postnatal Care in Ethiopia
Acronym: FPNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Addis Continental Institute of Public Health (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Della Berhanu, Research lead, Jhpiego
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00021096
Record Dates: First submitted 2022-08-30; First posted 2022-10-03 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Postnatal Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Women who agree to receive family led postnatal care (Experimental): This group will receive Family-led Postnatal Care-FPNC
  Interventions: Other: Family led postnatal care
- Women who receive standard of care for postnatal care (No Intervention): Women will get the standard of care for postnatal care

INTERVENTIONS:
Other: Family led postnatal care — Family-led Postnatal Care-FPNC A midwife involves families and uses a visual checklist to assess and counsel. The midwife then gives families the checklist and guides them how to retrieve a "home care kit" that has a blood pressure machine, infrared thermometer, and health education booklet.
  At home, families assess the health of postnatal mothers and newborns for 6 days, and then return the completed checklist and home care kit to the community location.
  Arms: Women who agree to receive family led postnatal care

SUMMARY:
Family-led Postnatal Care-FPNC A midwife involves families and uses a visual checklist to assess and counsel. The midwife then gives families the checklist along with information on how to retrieve a "homecare kit" that has a blood pressure machine, infrared thermometer, and health education booklet. At home, families assess the health of postnatal mothers and newborns for 6 days, and then return the completed checklist and homecare kit to the community location. A community health worker collects the checklists monthly. This study aims to assess the acceptability and feasibility of the FPNC and assess if FPNC increases the proportion of women/newborns who have a postnatal check in the first week after delivery and the proportion who seek care from a health provider when a postnatal danger sign is identified. The study will take approximately 12 months.

DETAILED DESCRIPTION:
Four health centers in Ada District of Oromia will be included in the study. Prior to FPNC introduction, the investigators will conduct a baseline survey over 8 weeks to measure coverage and content of postnatal checks on Days 3 and 7, as well as care-seeking behavior.

The health centers will then implement FPNC. Postnatal women, families, midwives, health extension workers, and homecare kit custodians will have the option to accept or decline participation in the study. At the end of the first- and second-months after FPNC implementation, the investigators will conduct qualitative interviews with mothers, families, midwives, health extension workers and homecare kit custodians.

Post intervention survey will take 8 weeks and will be conducted three months after FPNC is introduced. Coverage and content of postnatal checks in the first week will be abstracted weekly from FPNC checklists and care-seeking information will be collected through face-to-face interviews. The investigators will also conduct a quantitative measurement of sustainability of the FPNC intervention six months after the deadline through facility register data abstraction and review of completed checklists.

ELIGIBILITY:
Inclusion Criteria:

Health center discharge counselors

* Provides postnatal care at intervention health center
* Willing to participate in study

Postnatal women and family members

* Per participant report, age 15 years or older
* Delivered at the intervention health centers
* Maximum of Postnatal Day 1-3 at HC
* Intends to remain within catchment area for first week after birth
* Has family members who are willing to participate in the study
* Able and willing to provide consent

Husbands

* Per participant report, age 15 years or older
* Husband of eligible postnatal woman who has consented to participate
* Able and willing to provide consent

Family members

* Per participant report, age 15 years or older
* Family members of eligible postnatal women who have consented to participate
* Able and willing to provide consent

Health extension workers

* Works within catchment area of intervention health center
* Willing to participate in study

Home care custodians

* Able and willing to provide consent

Health facility managers

* Able and willing to provide consent

Exclusion Criteria:

Health center discharge counselors

* N/A

Postnatal women and family members

* Women who are unable to provide valid information because of mental or other serious health condition

Husbands

* N/A

Family members

* 15-18 year old members who are not emancipated minors (married or have children of their own)

Health extension workers

* Is not selected to participate (i.e., if there is more than one HEWs per health post)

Home care custodians

* N/A

Health facility managers

* N/A

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change in coverage (Mothers) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention (for approximately 8 weeks) and immediately after the intervention (for approximately 8 weeks), the investigators will measure the change in the proportion of postnatal women who have all three postnatal checks (within 1st day, 2nd-3rd days, and 4th-7th days).
Change in coverage (Newborns) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the proportion of newborns who have all three postnatal checks (within 1st day, 2nd-3rd days, and 4th-7th days).
Change in completeness (Mothers) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the proportion of postnatal women who had all specified PNC components assessed during all three postnatal checks (within 1st day, 2nd-3rd days, and 4th-7th days).
Change in completeness (Newborns) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the proportion of newborns who had all specified PNC components assessed during all three postnatal checks (within 1st day, 2nd-3rd days, and 4th-7th days).
Change in postnatal Contacts (Mothers) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the average number of PNC checks that are done for mothers in the first 7 days after delivery.
Change in postnatal Contacts (Newborns) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the average number of PNC checks that are done for newborns in the first 7 days after delivery.

SECONDARY OUTCOMES:
Change in Danger Sign Recognition (Mothers) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the proportion of postnatal women who had a postnatal danger sign identified in the first week after delivery.
  Proportion of newborns with a danger sign identified
  Proportion of women and newborns who seek care from a health provider when a postnatal danger sign is identified (disaggregated by type of provider and type of facility)
Change in Danger Sign Recognition (Newborns) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks).
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the proportion of newborns for whom a postnatal danger sign was identified in the first week after delivery.
Change in Care-Seeking (Mothers) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks)
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the proportion of postnatal women who sought care for an identified danger sign (disaggregated by type of provider and type of facility) in the first week after delivery.
Change in Care-Seeking (Newborns) | Pre-intervention (for approximately 8 weeks) and immediately after intervention (for approximately 8 weeks)
  Between pre-intervention and immediately after the intervention, the investigators will measure the change in the proportion of newborns for whom care was sought for an identified danger sign (disaggregated by type of provider and type of facility) in the first week after delivery.
Feasibility (Homecare Kit) | Immediately after the intervention (for approximately 8 weeks)
  Among postnatal women who are discharged from the facility after the intervention is initiated, the proportion whose family members retrieve the homecare kit. This will be part of the feasibility study.
Feasibility (Blood Pressure) | Immediately after the intervention (for approximately 8 weeks)
  Among postnatal women who are discharged from the facility after the intervention is initiated and those whose family retrieve the homecare kit, the proportion who report successful use of the blood pressure cuff. This will be part of the feasibility study.
Feasibility (Thermometer, Mothers) | Immediately after the intervention (for approximately 8 weeks)
  Among postnatal women who are discharged from the facility after the intervention is initiated and those whose family retrieve the homecare kit, the proportion who report successful use of the thermometer for themselves.
Feasibility (Thermometer, Newborns) | Immediately after the intervention (for approximately 8 weeks)
  Among postnatal women who are discharged from the facility after the intervention is initiated and those whose family retrieve the homecare kit, the proportion of who report successful use of the thermometer to check their newborn's health. This will be part of the feasibility study.
Feasibility (Communication) | Immediately after the intervention (for approximately 8 weeks)
  Among families who are discharged from the facility after the intervention is initiated and those whose family retrieve the homecare kit, the proportion who communicate with past homecare kit users. This will be part of the feasibility study.
Feasibility (Kit Return) | Immediately after the intervention (for approximately 8 weeks)
  Among families who are discharged from the facility after the intervention is initiated and those whose family retrieve the homecare kit, the proportion who return the homecare it by day 8. This will be part of the feasibility study.
Feasibility (Checklist Return) | Immediately after the intervention (for approximately 8 weeks)
  Among families who are discharged from the facility after the intervention is initiated and those whose family retrieve the homecare kit, the proportion who return the checklist to the custodian. This will be part of the feasibility study.
Feasibility (Checklist Collection) | Immediately after the intervention (for approximately 8 weeks)
  Among checklist brought to the homecare kit custodian, the proportion that are collected by the health extension workers. This will be part of the feasibility study.
Feasibility (Functional Kits) | Immediately after the intervention (for approximately 8 weeks)
  Among all the homecare kits distributed to custodians, the proportion that are 100% functional upon monthly checks of a random sample of homecare kits. This will be part of the feasibility study.
Feasibility (Register) | Immediately after the intervention (for approximately 8 weeks)
  Among all the homecare kit registers distributed to custodians, the proportion that are filled completely by the homecare kit custodian. This will be part of the feasibility study.
Acceptability (Checklist) | Immediately after the intervention (for approximately 8 weeks)
  Among postnatal women discharged from the facilities after the intervention is initiated, the proportion that accept a checklist form the discharge counselor. This will be part of the acceptability study.
Acceptability (Homecare Kit) | Immediately after the intervention (for approximately 8 weeks)
  Among postnatal women discharged from the facilities after the intervention is initiated and whose family retrieve the homecare kit, the proportion who report preferring the FPNC approach. This will be part of the acceptability study.
Acceptability (Perceptions of Discharge Counselors) | Immediately after the intervention (for approximately 8 weeks)
  Investigators will use qualitative methods to understand perceptions of discharge counselors on the acceptance and support for the FPNC approach. This will be part of the acceptability study.
Acceptability (Perceptions of Homecare Kit Custodians) | Immediately after the intervention (for approximately 8 weeks)
  Investigators will use qualitative methods to understand the homecare kit custodians' perceptions on the FPNC approach. This will be part of the acceptability study.
Acceptability (Perception of Health Managers) | Immediately after the intervention (for approximately 8 weeks)
  Investigators will use qualitative methods with health managers to understand their perceptions on the FPNC approach. This will be part of the acceptability study.
Acceptability (Perceptions of Health Extension Workers) | Immediately after the intervention (for approximately 8 weeks)
  Investigators will use qualitative methods with health extension workers to understand their perceptions on the FPNC approach. This will be part of the acceptability study.
Acceptability (Perceptions of Husbands and Family Members) | Immediately after the intervention (for approximately 8 weeks)
  Investigators will use qualitative methods with husbands and families to understand husbands' engagement in PNC. This will be part of the acceptability study.
Preference (Families') | Immediately after the intervention (for approximately 8 weeks)
  Among families that retrieve the homecare kit, the proportion that report a preference for the FPNC approach. This will address the area of values and preferences.
Satisfaction (Dsicharge counselors') | Immediately after the intervention (for approximately 8 weeks)
  The proportion of discharge counselors who report satisfaction with the FPNC approach, including discharge process. This will address the area of values and preferences.
Sustainability | Six months after the post-intervention survey.
  Among all the homecare kits distributed, the proportion that are functional at six months post intervention survey. This will be part of the sustainability assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Health centers in Ada Woreda, Bishoftu, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Per current Bill & Melinda Gates Foundation policy for study data